CLINICAL TRIAL: NCT05555082
Title: Can Massage During One Year Improve Health in Health-care Providers Working in Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Peter Johansson, Professor, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-01140
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Massage Therapy; Health-care Workers; Quality of Life; Psychological Distress
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: 50 health care professionals will receive massage monthly during 12 months. Massage will not be given during summer holiday. Thus, 30 minutes of massage will be given 10 times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massage (Experimental): 30 minutes of classical swedish massage given by a certified masseur 10 times monthly during 12 months
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — 10 times of 30 minutes Swedish classical Massage will be given monthly during one year. The massage will be give by a cerified masseur

SUMMARY:
The overall aim of this pilot study is to investigate the effect, "feasibility" and experiences of regular massage over 12 months on the mental and physical health of healthcare professionals, as well as the frequency of layoffs, sick leave and reported patient safety risk cases, as well as health economics

DETAILED DESCRIPTION:
A pilot and "feasibility" study with pre-post design. 50 health care professionals from the Medical Clinic, Vrinnevi Hospital in Norrköping are included. The participants perform 10 30 minute sessions of classic Swedish massage during 12 months by a certified masseur. Mental and physical health data is collected using questionnaires, blood and body weight. Data on layoffs, sick leave and patient safety risks are taken from the hospital's data register. Data regarding the participants' experience of receiving massages is collected during interviews.

ELIGIBILITY:
Inclusion Criteria:

Working at least for 50 % of fulltime

Main task working with patient care in the hospital ward

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johansson, Professor, Principal Investigator — Linköpings Universiet
Locations (2):
- Sweden (2):
  - Peter Johansson, Norrköping, Linköpings Universitet
  - Linkoping University, Norrköping

IPD SHARING:
Plan to Share IPD: No
At our university we have not yet any plan on how to deal with GDPR and sharing data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Massage
Started (25 patients started massage) | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Massage: Registered and assistant nurses working on a hospital ward received classic Swedish massage once per month for 12 months (about 10-12 sessions). Each 30-minute session used standard Swedish massage techniques-kneading, gliding, and tapping-focused on the back, shoulders, and neck to relieve work-related tension. Sessions were delivered by licensed therapists in a calm setting outside work hours, with the same therapist assigned to each participant. The study evaluated feasibility, including recruitment, adherence, satisfaction, and preliminary within-group effects on stress, mental health, sleep, pain, physical activity, work ability, and quality of life.
Arm/Group | Massage
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of smokers, ex-smokers and never smoked [Number; unit: Number of participants] — Self reported of smoking, or ex-smoker or never smoked
  Number of participants
    Smokers | 4
    Ex-smoker | 11
    Never smoked | 10

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Stress
Description: The Perceived Stress Scale-10 (PSS-10) is a 10-item self-report questionnaire measuring perceived stress during the past month. Total scores range from 0 to 40, with higher scores indicating greater perceived stress (i.e., worse outcome).
Time Frame: Baseline (start of massage) and 12 months (end of massage)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Massage
Number analyzed (Participants) | 25
units on a scale
  Basline | 17.4 (4.9)
  12 months | 13.9 (5.7)
Statistical Analysis 1: Comparison: Massage; Single-arm feasibility design; exploratory within-group analysis; Test type: Other — Single-arm feasibility design; exploratory within-group analysis; p = 0.021, Mixed Models Analysis — P-values reported for transparency; feasibility study not powered for hypothesis testing; Linear mixed model with repeated measures; maximum likelihood estimation; Mean Difference (Final Values) = -3.398, 95% CI 2-sided [-6.236 to -0.559] — Within-group change from baseline to 12 months
Statistical Analysis 2: Comparison: Massage; Test type: Other; Cohens d = 0.66

2. Secondary Outcome: Symptoms of Anxiety
Description: The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire assessing anxiety symptoms during the past two weeks. Each item is rated from 0 ("not at all") to 3 ("nearly every day"), giving a total score from 0 to 21. Higher scores indicate greater anxiety severity (worse outcome).
Time Frame: Baseline (start of massage and 12 months (end of massage).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Massage
Number analyzed (Participants) | 25
score on a scale
  Baseline | 6.8 (4.3)
  12 months | 5.5 (4.8)
Statistical Analysis 1: Comparison: Massage; "Single-arm feasibility design; exploratory within-group analysis; Test type: Other — Single-arm feasibility design; exploratory within-group analysis; p = 0.318, Mixed Models Analysis — P-values reported for transparency; study not powered for significance testing; Linear mixed model with repeated measures; maximum likelihood estimation; Median Difference (Final Values) = -1.328, 95% CI 2-sided [-4.013 to 1.357] — Within-group change from baseline to 12 months;
Statistical Analysis 2: Comparison: Massage; Test type: Other; Cohens d = 0.29

3. Secondary Outcome: Sleeping Problems
Description: The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia during the past two weeks. Scores range from 0 to 28, with higher scores indicating more severe insomnia.
Time Frame: ISI mean score from baseline (start of massage) to12 months (end of massage).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Massage
Number analyzed (Participants) | 25
score on a scale
  Baseline | 11.8 (4.6)
  12 months | 10.5 (6.6)
Statistical Analysis 1: Comparison: Massage; "Single-arm feasibility design; exploratory within-group analysis; Test type: Other — Single-arm feasibility design; exploratory within-group analysis; p = 0.28, Mixed Models Analysis — P-values reported for transparency; study not powered for significance testing; Linear mixed model with repeated measures; maximum likelihood estimation; Median Difference (Final Values) = -1.453, 95% CI 2-sided [-4.174 to 1.268] — Within-group change from baseline to 12 months
Statistical Analysis 2: Comparison: Massage; Test type: Other; Cohens d = 0.23

4. Secondary Outcome: Symptoms of Depression
Description: The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire assessing depressive symptoms during the past two weeks. Scores range from 0 to 27, with higher scores indicating greater depression severity.
Time Frame: PHQ-9 mean score from baseline (start of massage) to 12 months (end of massage).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Massage
Number analyzed (Participants) | 25
units on a scale
  Baseline | 7.2 (4.1)
  12-months | 4.9 (3.9)
Statistical Analysis 1: Comparison: Massage; "Single-arm feasibility design; exploratory within-group analysis; Test type: Other — Single-arm feasibility design; exploratory within-group analysis; p = 0.023, Mixed Models Analysis — P-values reported for transparency; study not powered for significance testing; Linear mixed model with repeated measures; maximum likelihood estimation; Median Difference (Final Values) = -2.122, 95% CI 2-sided [-3.917 to -0.326] — Within-group change from baseline to 12 months
Statistical Analysis 2: Comparison: Massage; Test type: Other; Cohens d = 0.57

5. Secondary Outcome: Health Related Quality of Life
Description: The RAND-36 Health Transition item asks respondents to rate their health compared with one year ago. Scores are transformed to a 0-100 scale. Higher scores indicate better perceived change (better outcome).
Time Frame: RAND-36 halth transition from baseline (start of massage) to 12 months (end of massage).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Massage
Number analyzed (Participants) | 25
score on a scale
  Baseline | 52 (23.5)
  12 months | 76.3 (26.9)
Statistical Analysis 1: Comparison: Massage; "Single-arm feasibility design; exploratory within-group analysis; Test type: Other — Single-arm feasibility design; exploratory within-group analysis; p = 0.004, Mixed Models Analysis — P-values reported for transparency; study not powered for significance testing; Linear mixed model with repeated measures; maximum likelihood estimation; Mean Difference (Final Values) = 24.876, 95% CI 2-sided [8.660 to 41.092] — Within-group change from baseline to 12 months
Statistical Analysis 2: Comparison: Massage; Test type: Other; Cohens d = 0.96

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Massage
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT05555082/Prot_SAP_000.pdf